CLINICAL TRIAL: NCT06177067
Title: A Phase 1 Study of Revumenib, Azacitidine, and Venetoclax in Pediatric and Young Adult Patients With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Study of Revumenib, Azacitidine, and Venetoclax in Pediatric and Young Adult Patients With Refractory or Relapsed Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAVAML; NCI-2023-10509 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Refractory Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia; Acute Leukemia of Ambiguous Lineage
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute | interventions — revumenib; venetoclax; Azacitidine; Drug Therapy; Methotrexate; Cytarabine

STUDY DESIGN:
Intervention Model Description: Participants with relapsed or refractory acute myeloid leukemia (AML) or acute leukemia of ambiguous lineage (ALAL) who meet the eligibility criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Eligible Participants (Experimental): All eligible patients receive the following intervention:
  Revumenib, Venetoclax, Azacitidine, Intrathecal chemotherapy
  Interventions: Drug: Revumenib; Drug: Venetoclax; Drug: Azacitidine; Drug: intrathecal (IT) chemotherapy; Drug: Cytarabine; Drug: Methotrexate

INTERVENTIONS:
Drug: Revumenib — Given by mouth (capsule or liquid solution) or liquid solution by Nasogastric tube (NG) or Gastrostomy tube (G-tube)
  Other Names: SNDX-5613
Drug: Venetoclax — Given by mouth (tablet) or by NG or G-tube
  Other Names: Venclextra®
Drug: Azacitidine — Given intravenously (IV) infusion
  Other Names: VIDAZA®; 5-azacitidine
Drug: intrathecal (IT) chemotherapy — Given intrathecal (IT)
  Other Names: ITMHA; methotrexate/hydrocortisone/cytarabine
Drug: Cytarabine — Given intrathecal (IT) as part of intrathecal (IT) chemotherapy.
  Other Names: Ara-C; Cytosar®
Drug: Methotrexate — Given intrathecal (IT) as part of intrathecal (IT) chemotherapy.
  Other Names: MTX; Trexall®

SUMMARY:
This is a research study to find out if adding a new study drug called revumenib to commonly used chemotherapy drugs is safe and if they have beneficial effects in treating patients with acute myeloid leukemia (AML) or acute leukemia of ambiguous lineage (ALAL) that did not go into remission after treatment (refractory) or has come back after treatment (relapsed), and to determine the total dose of the 3-drug combination of revumenib, azacitidine and venetoclax that can be given safely in participants also taking an anti-fungal drug.

Primary Objective

* To determine the safety and tolerability of revumenib + azacitidine + venetoclax in pediatric patients with relapsed or refractory AML or ALAL.

Secondary Objectives

* Describe the rates of complete remission (CR), complete remission with incomplete count recovery (CRi), and overall survival for patients treated with revumenib + azacitidine + venetoclax at the recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
Patients will receive revumenib + azacitidine + venetoclax in a dose-escalation fashion. The protocol starts at dose level 1. If there are no dose limiting toxicities at dose level 1, then patients will be treated at dose level 2, which equates to the dose of revumenib increasing from 65 to 95 mg/m^2 while the venetoclax exposure remains the same at 21 days. Alternatively, if there are dose limiting toxicities at dose level 1, then the dose level will be deescalated to dose level -1, which equates to the length of exposure of venetoclax being decreased from 21 days to 14 days, while the dose of revumenib stays at 65 mg/m^2. The doses of azacitidine will remain constant at all dose levels.

For patients whose primary physician considers that single agent revumenib is beneficial (e.g., transition to hematopoietic cell transplant), revumenib can be continued after discussing with study principal investigator. Patients who undergo HCT will be taken off therapy at the time of HCT, but will remain on study. Post-transplant therapy will be determined by the HCT physician.

Patients who do not go on to receive an HCT, may continue to receive revumenib, venetoclax and azacitidine as long as their primary physician considers it beneficial and there are no unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria: Participants must have a diagnosis of AML or ALAL and meet the criteria below:

* Refractory leukemia, defined as persistent leukemia after at least two courses of induction chemotherapy (one course for secondary AML), or relapsed leukemia, defined as the re-appearance of leukemia after the achievement of remission. Patients must have ≥5% blasts in the bone marrow as assessed by morphology or ≥1% blasts flow cytometry.

However, if an adequate bone marrow sample cannot be obtained (e.g., in a patient with acute megakaryoblastic leukemia with marrow fibrosis), patients may be enrolled if there is unequivocal evidence of leukemia with ≥5% blasts by morphology or ≥1% blasts flow cytometry in the blood.

* Presence of KMT2A rearrangement (KMT2Ar), NUP98 rearrangement (NUP98r), NPM1 mutation or fusion, PICALM::MLLT10, DEK::NUP214, UBTF-TD, KAT6A rearrangement (KAT6Ar), or SET::NUP214
* Adequate organ function, defined as total bilirubin < 1.5 × institutional upper limit of normal for age or normal conjugated bilirubin (for patients with known Gilbert's syndrome, total bilirubin <3 × the ULN) unless attributed to leukemia, calculated creatinine clearance ≥60 mL/min/1.73 m^2, and left ventricular ejection fraction ≥ 40%
* QTcF < 480 msec (average of triplicate)
* Age ≥ 1 year and ≤ 30 years. The upper age limit may be defined by each institution, but may not exceed 30 years.
* Lansky ≥ 60 for patients who are < 16 years old and Karnofsky ≥ 60% for patients who are > 16 years old.
* At least 14 days or 5 half-lives (whichever is longer) must have elapsed since the completion of myelosuppressive therapy, with the exception of low-dose therapy used for cytoreduction according to institutional standards, such as hydroxyurea or low-dose cytarabine (up to 200 mg/m^2/day). In addition, all toxicities must have resolved to grade 1 or less.
* Patients must have a leukocyte count <25,000 cells/uL. Low-dose therapy, such as hydroxyurea or cytarabine as described above, to achieve this limit is acceptable.
* For patients who have received prior HCT, there can be no evidence of GVHD and greater than 60 days must have elapsed since the HCT, and patients should be off calcineurin inhibitors for at least 28 days prior to the start of protocol therapy. Physiologic prednisone for the treatment of adrenal insufficiency is acceptable..
* Patients must be taking posaconazole or voriconazole, which must be started at least 24 hours prior to the start of therapy.
* Patients of reproductive potential must agree to use effective contraception for the duration of study participation.

Patients who meet the criteria listed above are eligible for enrollment and treatment on the trial. However, patients in first relapse who are suitable for and willing to receive intensive remission induction therapy should be offered such therapy if deemed appropriate by the treating physician.

Exclusion Criteria:

* Patients who are pregnant or breastfeeding are not eligible.
* Patients with Down syndrome, acute promyelocytic leukemia, juvenile myelomonocytic leukemia, or bone marrow failure syndromes are not eligible.
* Patients with uncontrolled infection are not eligible. Patients with infections that are controlled on concurrent anti-microbial agents are eligible.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of revumenib + azacitidine + venetoclax in pediatric patients with relapsed or refractory AML or ALAL | 43 days from the start of therapy.
  The primary endpoint is the recommended phase 2 dose (RP2D) of revumenib + azacitidine + venetoclax.

SECONDARY OUTCOMES:
The rates of complete remission (CR) | 43 days from the start of therapy
  CR is defined as bone marrow with < 5% blasts confirmed by flow cytometry, ANC ≥500/μL and platelets ≥50,000/μL without transfusions, and no evidence of extramedullary disease.
The rates of complete remission with incomplete count recovery (CRi) | 43 days from the start of therapy
  CRi is defined as bone marrow with <5% blasts confirmed by flow cytometry and ANC <500/μL or platelets <50,000/μL without transfusions
The overall survival of patients treated at the RP2D. | 1 year
  Kaplan-Meier estimates with 95% confidence intervals will be used to describe overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroto Inaba, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (9):
- United States (9):
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Mercy Hospital of Kansas City, Kansas City, Missouri
  - Memorial Sloan- Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern/Simmons Cancer Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols